CLINICAL TRIAL: NCT00510471
Title: A Phase 2 Multi-Center, Open-Label Study to Evaluate the Efficacy and Safety of Patient-Specific Immunotherapy, Recombinant Idiotype Conjugated to KLH (Id-KLH) and Administered With GM-CSF, in Patients With Follicular Non-Hodgkin's Lymphoma (fNHL) Following Primary Treatment With Rituximab and Chemotherapy (R-Chemo)
Brief Title: Personalized Active Immunotherapy (Vaccine Therapy) and Sargramostim Given After Standard of Care Treatment With Rituximab and Chemotherapy for Initial Treatment With Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Genitope Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2007-12
Record Dates: First submitted 2007-07-31; First posted 2007-08-02 (Estimated); Last update posted 2008-03-18 (Estimated); Status verified 2008-03

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

INTERVENTIONS:
Drug: autologous immunoglobulin idiotype-KLH conjugate vaccine

SUMMARY:
The treatment being investigated is a patient- and tumor-specific therapy known as a personalized active immunotherapy. Personalized active immunotherapy is an attempt to use a person's own immune system to combat disease. Sargramostim (a.k.a. GM-CSF) is given together with the personalized active immunotherapy because it may increase the immune system's response and, therefore, aid in the effect of the personalized active immunotherapy.

This approach has previously been studied in patients with follicular Non-Hodgkin's lymphoma and other B-cell malignancies. Encouraging efficacy results and a favorable safety profile have been seen to date in these studies.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Previously untreated follicular NHL
3. Stage III or IV disease requiring treatment
4. Able to receive rituximab and chemotherapy (rituximab with cyclophosphamide, vincristine, and prednisone either with or without doxorubicin)
5. Able to provide tumor sample adequate for Id-KLH manufacture
6. ≥ 18 years of age
7. At least one bi-dimensionally measurable lesion ≥ 2 cm by CT scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-05

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Keck School of Medicine of University Southern California, Los Angeles, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Indiana University Medical Center, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Weill Medical College of Cornell University, NY Presbyterian Hospital, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Providence Portland Cancer Center, Portland, Oregon

REFERENCES:
- See also: Click here for more information for untreated patients with follicular Non-Hodgkin's lymphoma who require treatment — http://www.genitope.com/